CLINICAL TRIAL: NCT01367600
Title: A Three-Month Open-Label Treatment Extension of Protocol MNTX 301
Brief Title: Open-Label Treatment Extension of Protocol MNTX 301
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Tage Ramakrishna, M.D., Progenics Pharmaceuticals, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MNTX 301EXT
Record Dates: First submitted 2011-05-27; First posted 2011-06-07 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Terminal Illness
Keywords: Advanced medical illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: SC Methylnaltrexone (MNTX)

INTERVENTIONS:
Drug: SC Methylnaltrexone (MNTX)

SUMMARY:
This study is an open-label extension allowing patients who have completed Protocol MNTX 301 to continue to receive SC MNTX.

ELIGIBILITY:
Inclusion Criteria:

1. Completion of protocol MNTX 301; Double-Blind Treatment and Open-Label Treatment
2. Negative pregnancy test

Exclusion Criteria:

1. Women who are pregnant and/or nursing
2. Any concurrent experimental drug therapy
3. Evidence of fecal impaction
4. Clinically significant active diverticular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2003-02; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | 3 months
  To provide access to continued treatment with MNTX administered SC, to patients who completed Progenics' MNTX 301.

SECONDARY OUTCOMES:
Change from baseline in pain scores | 3 months
  To provide access to continued treatment with MNTX administered SC, to patients who completed Progenics' MNTX 301.
Number of patients with opioid withdrawal symptoms | 3 months
  To provide access to continued treatment with MNTX administered SC, to patients who completed Progenics' MNTX 301.

CONTACTS AND LOCATIONS:
Overall Officials: Tage Ramakrishna, MD, Study Director — Progenics Pharmaceuticals, Inc.
Locations (1):
- Progenics Pharmaceuticals, Tarrytown, New York, United States